CLINICAL TRIAL: NCT06563076
Title: Evaluation of the Effectiveness of Vestibular Electrical Stimulation in Vestibular Rehabilitation
Brief Title: Effectiveness of Vestibular Electrical Stimulation in Vestibular Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Bilal Burak Bayraklı, Principal Investigator, Medical Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2-22-2962; 10026336 (Other: Ankara Bilkent City Hospital)
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Vestibular Diseases; Vestibular Disorder; Vestibular Vertigo
Keywords: Vertigo; Rehabilitation; TENS
MeSH Terms: conditions — Vestibular Diseases; Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation Group (Active Comparator): underwent vestibular rehabilitation program
  Interventions: Other: Vestibular Rehabilitation
- Vestibular Rehabilitation and Vestibular Electrical Stimulation Group (Active Comparator): underwent vestibular electrical stimulation (VES) in addition to the supervised vestibular rehabilitation program.
  Interventions: Other: Vestibular Rehabilitation; Other: Vestibular Electrical Stimulation

INTERVENTIONS:
Other: Vestibular Rehabilitation — supervised vestibular rehabilitation program
Other: Vestibular Electrical Stimulation — 80 Hz high frequency transcutaneous vestibular electrical stimulation (VES)
  Arms: Vestibular Rehabilitation and Vestibular Electrical Stimulation Group

SUMMARY:
This study aimed to evaluate the effectiveness of the vestibular rehabilitation program applied to patients with chronic unilateral vestibular hypofunction and the vestibular electrical stimulation applied to the trapezius muscles and cervical paravertebral muscles along with the rehabilitation program.

DETAILED DESCRIPTION:
This study included 40 patients with unilateral vestibular hypofunction findings, aged between 18 and 65, and whose unilateral vestibulo-ocular reflex (VOR) gain for any semicircular canal was below 0.7 based on the video head impulse test (vHIT) test, were randomized into two groups. While one group underwent a supervised vestibular rehabilitation program for 4 weeks, the other group received 80 Hz high frequency transcutaneous vestibular electrical stimulation (VES) in addition to the supervised vestibular rehabilitation program. The treatment was applied to each group, 3 days a week, for a total of 12 sessions. Detailed musculoskeletal system examinations and vestibular system examinations of the included patients were performed, and sociodemographic characteristics (age, gender, body mass index (BMI), education level) were recorded. Both groups were tested before treatment and at the end of the 4th week, Dizziness Disability Inventory (DHI), Visual Analogue Scale (VAS), Berg Balance Scale (BBS), Timed Up and Go Test (TUG), Activity-Specific Balance and Confidence Scale (ABCs), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI) and Static Posturography.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Patients who were evaluated by a Neurologist, Physical Medicine and Rehabilitation Specialist and otorhinolaryngologist and diagnosed with chronic unilateral vestibular hypofunction and have findings of chronic unilateral vestibular hypofunction
* Patients whose VOR gain for any unilateral semicircular canal based on vHIT test is below 0.7
* Patients who volunteered to participate in the study and signed the consent forms

Exclusion Criteria:

* Existing neurological or mental disorders
* Patients using vestibulosuppressant drugs
* Stroke, head trauma and other neurological diseases
* Patients with a history of brain surgery
* Patients with severely limited neck joint range of motion (those with a limitation of 45 degrees or more)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | Baseline and after 4 weeks
  'Dizziness Handicap Inventory (DHI)' consists of 25 items that determine the functional and sensory consequences of vestibular system diseases as well as the factors that aggravate dizziness and balance disorders.
  Questions 1, 4, 8, 11, 13, 17 and 25 of the scale are structured to measure physical disability; questions 2, 9, 10, 15, 18, 20, 21, 22 and 23 are structured to measure emotional disability; questions 3, 5, 6, 7, 12, 14, 16, 19 and 24 are structured to measure functional disability. Each question is scored as yes (4 points), no (0 points) and sometimes (2 points). The level of disability can be categorized according to the scale: 16-34 points = mild disability; 36-52 points = moderate disability; 54+ points = severe disability

SECONDARY OUTCOMES:
Dizziness Severity Visual Analog Scale | Baseline and after 4 weeks
  Dizziness Severity: Using the Visual Analog Scale (VAS), patients are asked to indicate the severity of dizziness they have felt in the last week on a 10-centimeter chart. 0: no symptoms, 10: symptoms are evaluated as very severe.
Timed Up and Go Test | Baseline and after 4 weeks
  Functional mobility and fall risk in patients are assessed with a timed up and go test. Patients were asked to get up from a standard arm chair, walk a distance of three meters, come back and sit down, and the time was calculated in seconds. When the timed up and go test is completed in more than 12 seconds, the risk of falling is considered to be increased.
Berg Balance Score | Baseline and after 4 weeks
  The "Berg Balance Scale" is used to determine the risk of falling in patients. It is a scale that shows whether patients can maintain their balance while performing 14 different tasks. It includes tasks such as sitting without support, standing up without support, standing in tandem, sitting down while standing, picking up objects from the floor, looking back while standing, standing on one leg, standing with eyes closed. Scoring is between 0 (cannot do) and 4 (safely do). The maximum score is 56.
Activity Specific Balance and Confidence Scale | Baseline and after 4 weeks
  The confidence that patients feel during their daily living activities at home and in the community is assessed with the "Activity Specific Balance and Confidence Scale (ABC)". It consists of 16 questions and each question is given a score between 0 (I have no confidence) and 100 (I have full confidence). All scores are added up and divided by 16 to obtain the main score. The risk of falling increases at 67 points and below. Home dependency increases at 50 points and below. A score between 50 and 80 indicates moderate limitation, and a score of 80 and above indicates community activity.
Beck Depression Inventory | Baseline and after 4 weeks
  The Beck Depression Inventory is used to identify the risk of depression in adults and to measure changes in the severity and level of depression symptoms. It consists of 21 questions about depression symptoms, two about emotions, eleven about cognitive symptoms, two about behaviors, five about physical symptoms, and one about interpersonal symptoms. Each question is scored from 0 to 3, resulting in a total score of 0 to 63.
Beck Anxiety Inventory | Baseline and after 4 weeks
  It is designed to measure the severity of anxiety symptoms experienced by individuals. Subjective anxiety and physical symptoms are questioned. It is a self-report scale consisting of 21 items and scored between 0 and 3 based on a Likert scale. The total score ranges from 0 to 63. Higher total scores indicate more severe levels of anxiety experienced by the individual.
Static Posturography | Baseline and after 4 weeks
  The ''Limits of Stability'' (LOS) test, which measures the maximum limit at which people can stand in order to remain stable in order to maintain balance when leaning in certain directions, is evaluated with the Hur Smart Balance Static Posturography device. This protocol is used to test the stability limits of the person in four directions. The tested person stands in the positions of leaning forward, leaning back, leaning left and leaning right, respectively, from the normal standing position. As a result of the measurements, the LOS values of each evaluation are recorded by the device.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Burak Bayraklı, M.D, Principal Investigator — Ankara City Hospital Bilkent; Ömer Kuzu, M.D, Study Chair — Ankara City Hospital Bilkent; Canan Çelik, Professor, Study Director — Ankara City Hospital Bilkent; Özlem Öztürk Tan, M.D, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No